CLINICAL TRIAL: NCT00265980
Title: Leptin in Human Energy and Neuroendocrine Homeostasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by sponsor. Lack of funding.
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AAAA5988; R01DK064773 (NIH)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Weight Loss
Keywords: Leptin; Obesity; Energy; Autonomics; Neuroendocrine
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Sodium Chloride; Leptin; metreleptin

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, crossover study: half of the subjects had placebo first and half had leptin first. The order does not affect data analysis.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Weight initial (No Intervention): Subjects undergo studies at their usual body weight which is used as a baseline against which to compare subjects following weight loss with or without leptin repletion.
- Weight -10% placebo (Placebo Comparator): Subjects are studied while at a 10% reduced body weight and receiving placebo injections for 5 weeks.
  Interventions: Drug: Subcutaneous Placebo
- Weight -10% leptin (Experimental): Subjects are studied while at a 10% reduced body weight and receiving leptin injections for 5 weeks.
  Interventions: Drug: Leptin

INTERVENTIONS:
Drug: Subcutaneous Placebo — Twice daily injections of saline in the same volume as will be used for leptin injections.
  Other Names: Saline
  Arms: Weight -10% placebo
Drug: Leptin — Leptin will be given as twice daily subcutaneous injections in doses titrated to replicate 8 a.m. circulating leptin concentrations measured in the same subjects prior to weight loss.
  Other Names: Metreleptin
  Arms: Weight -10% leptin

SUMMARY:
Previous work in our laboratory, and many others, has shown that body weight is regulated. When anyone, fat or thin, tries to maintain a reduced body weight, many systems affecting energy balance (skeletal muscle, neuroendocrine, and autonomic systems) conspire to slow metabolic rate thus favoring the regain of lost weight. Individuals with leptin deficiency are remarkably similar to weight-reduced individuals. Their metabolism, thyroid hormones, and sympathetic nervous system activity are all low despite their obesity. While administration of leptin to leptin-deficient humans results in substantial weight loss and increases in energy expenditure. However, leptin administration to leptin-sufficient humans at usual body weight has little or no effect on weight unless given in doses 10-20 times what would be considered to be in the normal physiological range. This study examines the hypothesis that leptin is "read" by various systems regulating energy balance as an indicator of how much energy we have stored and that the body perceives the weight-reduced state as a condition of relative leptin insufficiency. Within this model, restoration of leptin to levels present prior to weight loss should relieve much of the metabolic opposition to keeping weight off. Preliminary studies support this hypothesis.

DETAILED DESCRIPTION:
The failure of obesity treatments to sustain weight reduction is widely recognized. The central hypotheses of these studies are that: 1) Energy and neuroendocrine homeostatic systems are altered during the maintenance of a reduced body weight in a manner that favors weight regain; 2) These changes occur because weight-reduced individuals are in a state of relative leptin deficiency due to loss of body fat; and 3) Therefore these changes accompanying the maintenance of a reduced body weight will be reversed if circulating leptin concentrations are restored to those that were present prior to weight reduction. Maintenance of a reduced body weight is associated with integrated autonomic and neuroendocrine changes that reduce energy expenditure and increase food intake in a manner that is similar to that seen in rodents and humans who are deficient in, or resistant to, the adipocyte-derived hormone leptin.

Systemic leptin administration to leptin-deficient rodents and humans reverses the metabolic (hypometabolism, hyperphagia), autonomic (increased parasympathetic and decreased sympathetic nervous system tone), and neuroendocrine changes that characterize the leptin-deficient state. The proposed studies focus on the neuroendocrine, autonomic, and metabolic changes that characterize the reduced-obese individual, and the effects on these phenotypes of restoration of circulating concentrations of leptin to levels present prior to weight loss.

Healthy lean and overweight subjects are admitted to the General Clinical Research Center at Columbia University Medical College and placed on a liquid formula diet. Calories are adjusted until weight is stable and then subjects undergo testing of neuroendocrine, autonomic, and metabolic function. All subjects undergo an in-patient 10% weight reduction. Subjects are studied in a single blind placebo control design in which they are studied at usual weight and while maintaining a 10% reduced weight. At either usual weight or reduced state subjects undergo a single blind crossover placebo/control study in which they receive placebo, leptin injections while on an isocaloric diet either at usual weight or following a 10% weight loss.

During each of these study periods, subjects will undergo detailed evaluation of 1) energy expenditure; 2) autonomic nervous system tone (serial blockade of sympathetic and parasympathetic inputs, heart rate variability analyses, and urinary catecholamine excretion); 3) hypothalamic-pituitary-thyroid, -adrenal and -gonadal, axis function; 4) adipose tissue gene expression; 5) other molecules (e.g., adiponectin, ghrelin, PYY) that may influence neuroendocrine and metabolic function. The results of these studies will further delineate the physiology of body weight regulation and of leptin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy lean or overweight males and females who have sustained their current weight for at least 6 months.

Exclusion Criteria:

* Pregnancy
* Any illness or chronic medication that affect energy expenditure, neuroendocrine function, autonomic function or that would impair ability to tolerate a prolonged hospital stay including rapid weight reduction and vigorous exercise.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2002-07 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rosenbaum, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Background] Rosenbaum M, Goldsmith R, Bloomfield D, Magnano A, Weimer L, Heymsfield S, Gallagher D, Mayer L, Murphy E, Leibel RL. Low-dose leptin reverses skeletal muscle, autonomic, and neuroendocrine adaptations to maintenance of reduced weight. J Clin Invest. 2005 Dec;115(12):3579-86. doi: 10.1172/JCI25977. PMID 16322796
- [Background] Rosenbaum M, Murphy EM, Heymsfield SB, Matthews DE, Leibel RL. Low dose leptin administration reverses effects of sustained weight-reduction on energy expenditure and circulating concentrations of thyroid hormones. J Clin Endocrinol Metab. 2002 May;87(5):2391-4. doi: 10.1210/jcem.87.5.8628. PMID 11994393
- [Background] Baldwin KM, Joanisse DR, Haddad F, Goldsmith RL, Gallagher D, Pavlovich KH, Shamoon EL, Leibel RL, Rosenbaum M. Effects of weight loss and leptin on skeletal muscle in human subjects. Am J Physiol Regul Integr Comp Physiol. 2011 Nov;301(5):R1259-66. doi: 10.1152/ajpregu.00397.2011. Epub 2011 Sep 14. PMID 21917907
- [Background] Hinkle W, Cordell M, Leibel R, Rosenbaum M, Hirsch J. Effects of reduced weight maintenance and leptin repletion on functional connectivity of the hypothalamus in obese humans. PLoS One. 2013;8(3):e59114. doi: 10.1371/journal.pone.0059114. Epub 2013 Mar 21. PMID 23555620
- [Background] Rosenbaum M, Leibel RL. 20 years of leptin: role of leptin in energy homeostasis in humans. J Endocrinol. 2014 Oct;223(1):T83-96. doi: 10.1530/JOE-14-0358. Epub 2014 Jul 25. PMID 25063755
- [Background] Page-Wilson G, Reitman-Ivashkov E, Meece K, White A, Rosenbaum M, Smiley RM, Wardlaw SL. Cerebrospinal fluid levels of leptin, proopiomelanocortin, and agouti-related protein in human pregnancy: evidence for leptin resistance. J Clin Endocrinol Metab. 2013 Jan;98(1):264-71. doi: 10.1210/jc.2012-2309. Epub 2012 Nov 1. PMID 23118421
- [Background] Kissileff HR, Thornton JC, Torres MI, Pavlovich K, Mayer LS, Kalari V, Leibel RL, Rosenbaum M. Leptin reverses declines in satiation in weight-reduced obese humans. Am J Clin Nutr. 2012 Feb;95(2):309-17. doi: 10.3945/ajcn.111.012385. Epub 2012 Jan 11. PMID 22237063
- [Result] Rosenbaum M, Goldsmith RL, Haddad F, Baldwin KM, Smiley R, Gallagher D, Leibel RL. Triiodothyronine and leptin repletion in humans similarly reverse weight-loss-induced changes in skeletal muscle. Am J Physiol Endocrinol Metab. 2018 Nov 1;315(5):E771-E779. doi: 10.1152/ajpendo.00116.2018. Epub 2018 Jun 19. PMID 29920214

RESULTS

PARTICIPANT FLOW:
Groups:
- Leptin Depletion Study Participants (Total): Each of the 22 participant went through the stages (arms) of obtaining the initial weight (Weight Initial), reducing weight maintenance (placebo injection), and repletion of leptin (leptin injection).
Period: Overall Study
Arm/Group | Leptin Depletion Study Participants (Total)
Started | 22
Weight Initial | 22
Weight -10% Placebo | 22
Weight -10% Leptin | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Leptin Depletion Study Participants (Total)
Number analyzed (Participants) | 22
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 34.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 22
Fa-free mass (FFM) [Mean (Standard Deviation); unit: kg] | 62.4 (14.3)

OUTCOME MEASURES:

1. Primary Outcome: Total Energy Expenditure (TEE)
Description: To measure the metabolic changes associated with maintenance of a reduced body weight (in kcal/day)
Time Frame: Baseline, 11 weeks, 18 weeks
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Leptin Depletion Study Participants (Total)
Number analyzed (Participants) | 22
kcal/day
  Weight initial | 3131 (500)
  Weight -10% placebo | 2457 (410)
  Weight -10% leptin | 2766 (799)

2. Secondary Outcome: TEE/FFM
Description: To measure the total energy expenditure/fat-free mass (FFM) (in kcal/kg).
Time Frame: Baseline, 11 weeks, 18 weeks
Measure: Mean (Standard Deviation); unit: kcal/kg
Arm/Group | Leptin Depletion Study Participants (Total)
Number analyzed (Participants) | 22
kcal/kg
  Weight initial | 51.1 (6.3)
  Weight -10% placebo | 41.7 (6.2)
  Weight -10% leptin | 48.1 (12.7)

ADVERSE EVENTS:
Time Frame: 18 weeks
Groups:
- Leptin Depletion Study Participants (Total): Each of the 22 participant went through the stages of obtaining the initial weight (Weight Initial), reducing weight maintenance (placebo injection), and repletion of leptin (leptin injection). Since adverse events are not the primary focus of this study, the events were not collected and analyzed by the stages but for each participant during the entire study participation, therefore the data is combined.
Arm/Group | Leptin Depletion Study Participants (Total)
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes